CLINICAL TRIAL: NCT07277920
Title: Evaluation of Reflectance Confocal Microscopy (RCM) Features in Surgically Excised Atypical Melanocytic Lesions and Their Correlation With Next-Generation Sequencing (NGS) Patterns
Brief Title: Reflectance Confocal Microscopy and Molecular Correlation in Atypical Melanocytic Lesions
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Francesca Farnetani, Professor / PI, University of Modena and Reggio Emilia
Other Study IDs: UNIMORE-DERM-2025-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Melanocytic Nevi; Melanoma (Skin Cancer); Next Generation Sequencing (NGS)
MeSH Terms: conditions — Nevus, Pigmented; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational, prospective cohort study aims to evaluate the diagnostic relevance of Reflectance Confocal Microscopy (RCM) features in atypical melanocytic lesions scheduled for surgical excision, and to correlate these imaging features with molecular profiles obtained through Next-Generation Sequencing (NGS). Approximately 200 consecutive lesions, including atypical nevi and early-stage melanomas, will be analyzed from patients attending the Videomicroscopy and Confocal Clinic at the Dermatology Department of the University Hospital of Modena.

The primary objective is to assess the diagnostic significance of RCM features-specifically atypical cells and disarrangement of the dermoepidermal junction (DEJ)-for early detection of melanoma. Secondary objectives include correlating RCM morphological patterns with NGS-derived genetic alterations and identifying molecular signatures that differentiate early-stage melanomas from benign nevi.

All procedures are performed as part of routine clinical care, including dermoscopic and confocal evaluation, surgical excision, histopathology, and molecular analysis on formalin-fixed, paraffin-embedded blocks. Data will be anonymized, securely stored, and analyzed to determine associations between imaging and genetic variables. This study integrates morphological and molecular data to refine diagnostic workflows and improve early melanoma detection.

DETAILED DESCRIPTION:
Background and Rationale

Reflectance confocal microscopy (RCM) is a non-invasive imaging technique that allows in vivo evaluation of the skin with near-histologic resolution. Integrating RCM into clinical dermatology has been shown to reduce unnecessary excisions of benign lesions and improve diagnostic accuracy compared with dermoscopy alone.

Next-Generation Sequencing (NGS) enables the identification of key genetic mutations in atypical nevi and melanomas, providing valuable insights into their biological behavior and potential malignant transformation.

This study aims to evaluate the correlation between characteristic RCM features and molecular findings obtained through NGS in melanocytic lesions already scheduled for surgical excision, to improve early diagnosis of melanoma and risk classification.

Objectives Primary Objective

To assess the diagnostic relevance of characteristic RCM features - specifically atypical cells and DEJ disarrangement - in melanocytic lesions already scheduled for surgical excision due to dermoscopic suspicion of atypical nevus or melanoma.

Secondary Objectives

To correlate RCM morphological features with molecular profiles obtained through NGS in both nevi and early-stage melanomas, comparing the genetic and morphologic patterns between these two groups.

To identify distinctive biological and molecular signatures that may differentiate early-stage melanomas from benign nevi, providing potential markers for early diagnosis and risk stratification.

Funding Statement

This study is funded by the European Union - NextGenerationEU, through the Italian Ministry of University and Research (MUR) under PNRR - M4C2-I1.3 Project PE_00000019 HEAL ITALIA, CUP E93C22001860006.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of cutaneous lesions with dermoscopic and reflectance confocal microscopy suspicion of melanocytic neoplasia, already scheduled for surgical excision
* Written informed consent obtained

Exclusion Criteria:

* Age < 18 years
* Lesions not scheduled for excision or with uncertain dermoscopic diagnosis
* Lack of informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 200 melanocytic lesions from adult patients (age ≥18 years) scheduled for surgical excision due to dermoscopic suspicion of atypical nevus or early-stage melanoma will be included. Patients of all genders are eligible. Lesions will be evaluated using routine clinical assessment, dermoscopy, and Reflectance Confocal Microscopy (RCM). Histopathological evaluation will be performed on all excised lesions. Molecular analysis via Next-Generation Sequencing (NGS) will be performed on lesions with available tissue, and not all lesions may undergo NGS. Participants are recruited consecutively at the Videomicroscopy and Confocal Clinic, Dermatology Department, University Hospital of Modena.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic relevance of RCM features in atypical melanocytic lesions | through study completion, an average of 1 year
  Evaluation of the presence of atypical cells (>20 µm, dendritic or round, suprabasal or at the dermoepidermal junction level) and disarrangement of the dermoepidermal junction (non-edged papillae, chaotic patterns, architectural irregularity) using Reflectance Confocal Microscopy (RCM), and comparison with histopathological diagnosis.

SECONDARY OUTCOMES:
Differential gene expression profiles distinguishing nevi and early-stage melanomas | through study completion, an average of 1 year
  Quantitative assessment of molecular features obtained through genomic/molecular analysis to identify patterns that distinguish benign nevi from early-stage melanomas. Data will be summarized as differential expression levels and/or frequency of molecular alterations.

OTHER OUTCOMES:
Correlation between RCM morphological patterns and NGS-derived molecular signatures | through study completion, an average of 1 year
  Outcome Measure Description
  Quantitative correlation analysis between:
  RCM morphological features, measured using Reflectance Confocal Microscopy (RCM) (e.g., presence of atypical cells, dermoepidermal junction disarrangement, architectural irregularity), summarized as categorical imaging features, and
  NGS-derived molecular signatures, measured through Next-Generation Sequencing (NGS), including identification of specific genes showing differential expression or genomic alterations, not only presence/absence of alterations.
  The reported outcome will be the correlation coefficient between imaging-defined RCM patterns and gene-level molecular profiles identified through NGS.
  Unit of Measure:
  Correlation coefficient (r value)
  Measurement Tools:
  Reflectance Confocal Microscopy (RCM) for morphological features
  Next-Generation Sequencing (NGS) for molecular signatures

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Department, University Hospital of Modena, Modena, Mo, Italy

REFERENCES:
- [Background] Mesbah Ardakani N. Dysplastic/Clark naevus in the era of molecular pathology. Australas J Dermatol. 2019 Aug;60(3):186-191. doi: 10.1111/ajd.13019. Epub 2019 Mar 10. PMID 30854639
- [Background] Piepkorn MW, Barnhill RL, Elder DE, Knezevich SR, Carney PA, Reisch LM, Elmore JG. The MPATH-Dx reporting schema for melanocytic proliferations and melanoma. J Am Acad Dermatol. 2014 Jan;70(1):131-41. doi: 10.1016/j.jaad.2013.07.027. Epub 2013 Oct 28. PMID 24176521
- [Background] Ferrara G, Argenziano G, Soyer HP, Corona R, Sera F, Brunetti B, Cerroni L, Chimenti S, El Shabrawi-Caelen L, Ferrari A, Hofmann-Wellenhof R, Kaddu S, Piccolo D, Scalvenzi M, Staibano S, Wolf IH, De Rosa G. Dermoscopic and histopathologic diagnosis of equivocal melanocytic skin lesions: an interdisciplinary study on 107 cases. Cancer. 2002 Sep 1;95(5):1094-100. doi: 10.1002/cncr.10768. PMID 12209696
- [Background] Kozubek J, Ma Z, Fleming E, Duggan T, Wu R, Shin DG, Dadras SS. In-depth characterization of microRNA transcriptome in melanoma. PLoS One. 2013 Sep 4;8(9):e72699. doi: 10.1371/journal.pone.0072699. eCollection 2013. PMID 24023765
- [Background] Sadrolashrafi K, Cotter DG. Not Your Mother's Melanoma: Causes and Effects of Early Melanoma Diagnosis. Dermatopathology (Basel). 2022 Nov 27;9(4):368-378. doi: 10.3390/dermatopathology9040043. PMID 36547217
- [Background] Navarrete-Dechent C, DeRosa AP, Longo C, Liopyris K, Oliviero M, Rabinovitz H, Marghoob AA, Halpern AC, Pellacani G, Scope A, Jain M. Reflectance confocal microscopy terminology glossary for nonmelanocytic skin lesions: A systematic review. J Am Acad Dermatol. 2019 May;80(5):1414-1427.e3. doi: 10.1016/j.jaad.2018.12.007. Epub 2018 Dec 8. PMID 30529706
- [Background] Pellacani G, Farnetani F, Gonzalez S, Longo C, Cesinaro AM, Casari A, Beretti F, Seidenari S, Gill M. In vivo confocal microscopy for detection and grading of dysplastic nevi: a pilot study. J Am Acad Dermatol. 2012 Mar;66(3):e109-21. doi: 10.1016/j.jaad.2011.05.017. Epub 2011 Jul 13. PMID 21742408
- [Background] Argenziano G, Catricala C, Ardigo M, Buccini P, De Simone P, Eibenschutz L, Ferrari A, Mariani G, Silipo V, Sperduti I, Zalaudek I. Seven-point checklist of dermoscopy revisited. Br J Dermatol. 2011 Apr;164(4):785-90. doi: 10.1111/j.1365-2133.2010.10194.x. Epub 2011 Mar 10. PMID 21175563
- [Background] Alma A, Beretti F, Bonilauri C, Chester J, Kaleci S, Ciardo S, Bertoni L, Pellacani G, Farnetani F. Atypical naevi in dermoscopy and reflectance confocal microscopy: correlation between immunohistochemistry and diagnostic patterns of atypia. Clin Exp Dermatol. 2024 Dec 23;50(1):172-174. doi: 10.1093/ced/llae326. No abstract available. PMID 39180293
- [Background] Gandini S, Sera F, Cattaruzza MS, Pasquini P, Abeni D, Boyle P, Melchi CF. Meta-analysis of risk factors for cutaneous melanoma: I. Common and atypical naevi. Eur J Cancer. 2005 Jan;41(1):28-44. doi: 10.1016/j.ejca.2004.10.015. PMID 15617989